CLINICAL TRIAL: NCT04115813
Title: Transitioning Adolescents to HIV Self-Management in Zambia (Known as: Project YES: Youth Engaging for Success)
Brief Title: Project YES! Youth Engaging for Success
Acronym: Project YES!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Population Council (Other); Arthur Davison Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00007870
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: HIV/AIDS
Keywords: Adolescents; Young Adults; Antiretroviral Therapy; Caregivers; Support Groups
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: After about 6 months and the completion of the initial intervention the intervention arm went into a less intensive maintenance phase and the comparison arm started to receive the intervention.
Who Masked: Outcomes Assessor
Masking Description: The laboratory staff testing the HIV blood for viral load levels were masked to the participants randomized allocation to the intervention or comparison arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention arm participants received the Project YES! intervention for the first phase and then after midline data collection went into a maintenance phase.
  Interventions: Behavioral: Project YES! Youth Engaging for Success
- Comparison Arm (Other): The comparison arm was a usual care arm during the first phase (and primary analysis). After midline data collection the comparison arm began receiving the Project YES! intervention.
  Interventions: Behavioral: Project YES! Youth Engaging for Success

INTERVENTIONS:
Behavioral: Project YES! Youth Engaging for Success — Participants in the intervention were offered once a month one-on-one meetings and group meetings with their assigned youth peer mentors over approximately six months. The participant's caregiver could also attend up to 3 caregiver support groups held at the clinic (every other month). In addition, intervention participants in the children's hospital were assessed (clinical and psycho social factors) for physical transition to an adult clinic. After midline data collection, the intervention arm went into a maintenance phase, meeting with the youth peer mentor every other month (3 times). Participants in the comparison arm after midline started the Project YES! intervention as described above. Primary analysis was conducted using midline data.

SUMMARY:
Youth-led strategies remain untested in clinic-based programs to achieve viral suppression (VS) and reduce self-stigma (feelings of worthlessness/shame) among adolescents and young adults (AYA) living with HIV in sub-Saharan Africa. In response, Project YES! will conduct a randomized controlled trial to test the impact of a theory-based intervention that places trained and paid HIV-positive youth peer mentors (YPMs) in four HIV clinics in Ndola, Zambia. AYA, ages 15 to 24 years, will be randomly assigned to either an intervention arm, consisting of monthly one-on-one and small group sessions with a YPM and optional caregiver support groups, or a usual care arm. Survey data and blood samples will be collected and analyzed to test the hypothesis that youth who are in the intervention group will experience more viral suppression than youth in the comparison group.

DETAILED DESCRIPTION:
BACKGROUND/INTRODUCTION While the literature on pediatric chronic illnesses often emphasizes the needs of adolescents transitioning from pediatric to adult care, there is no published literature on interventions to support HIV-positive adolescents transitioning to adult care and/or HIV self-management in sub-Saharan Africa (SSA). Similarly, there is virtually no data on how to best engage families and peers to support youth (YLHIV) with their care needs in SSA, despite the known impact families and peers have on adolescent health. For example, a 2015 review found only 14 studies on adolescents living with HIV (ALHIV) transitioning to adult care, all of which were conducted in the US or UK and the majority of which were qualitative studies with sample sizes of 50 participants or fewer. A 2016 systematic review examined the literature to assess the effectiveness of self-management interventions for young people across chronic illnesses. Out of 42 randomized controlled trials included in the review, none were conducted in SSA. The authors note that most interventions focused on the medical aspects of self-management rather than psycho-social issues. The authors also discuss the potential role for online peer support. These findings correspond with other articles that define three specific aspects of self-management: medical management (e.g., treatment adherence), role management (e.g., social participation), and emotional or identity management (e.g., feelings, stigma).

Despite this lack of evidence on how to support youth, the need remains great. Preliminary analysis of routine viral load (VL) testing conducted among ALHIV clinic attendees at the Arthur Davison Children's Hospital (ADCH) in Ndola, Zambia revealed that around 50% of ALHIV have viral failure defined as 1000 copies/ml or higher. This staggering percentage underscores the urgent need for assistance with care for this population.

This study will address this gap by testing a peer-mentoring program to implement the AIDS Support & Technical Assistance Resources (AIDSTAR-One) toolkit for transition (https://aidsfree.usaid.gov/sites/default/files/final_alhivtoolkit_web.pdf). AIDSTAR-One developed this toolkit as a resource for health care providers to support youth transitioning to HIV self-management as well as their caregivers. The current version, released in 2014, includes a transition readiness checklist designed for health care providers to monitor an adolescent's ability to self-manage his/her HIV. The toolkit also has corresponding modules that cover 10 subject areas deemed critical for youth's successful HIV self-management, including psychosocial development, mental health, sexual and reproductive health, alcohol and substance abuse, beneficial disclosure and clinical considerations.

While there have been no large scale implementations of this toolkit, the initial version was piloted in Kenya in 2012 "to inform final adaptations prior to dissemination" A survey conducted among 17 health care and community care providers in Kenya who were trained on the AIDSTAR-One toolkit, found that a majority were satisfied with the kit. A key concern expressed, however, was the time needed to implement the toolkit approach in settings where providers are overburdened. A subsequent key recommendation made by providers during this pilot evaluation was to expand the use of the toolkit to community-based providers, including specifically peer counselors or mentors. Peer mentors, especially those who are trained well and given paid positions, have been effective in other settings, such as the Mothers to Mothers program in South Africa r the Restless Development program in Zambia. In South Africa, paid mentors who are mothers themselves and had undergone prevention of mother to child HIV transmission (PMTCT) learned concrete employable skills and were integrated into the health care system to mentor women undergoing PMTCT. In Zambia, a youth intervention was conducted that placed young adults (18 to 24 years) in government schools to teach a Ministry of Education life skills course. Again, these youth mentors were paid, well trained, and given a position within the system. Results from an evaluation found that students in the schools with youth mentors had more HIV and reproductive health knowledge, and lower levels of stigma and sexual risk-taking behaviors, than their peers in schools without youth mentors. In this study, peer mentors will be integrated into the health care system to implement the toolkit.

This study will further explore the potential integration of violence-related content into the intervention. Despite limited existing literature on violence victimization among HIV-positive youth in SSA, studies among adults in SSA and elsewhere have documented negative impacts of violence victimization on HIV disclosure, linkage to care, and engagement and retention in care. A deeper understanding is needed of the types of violence experienced by youth, the influence of such violence on youth's HIV care and treatment, and the potential role of the adapted AIDSTAR-One toolkit for transition in addressing such violence.

STUDY GOAL AND AIMS

The overall goal of this study is to test a peer-mentoring approach to implementing the AIDSTAR-One toolkit to improve HIV-related outcomes, including viral suppression, among youth as they transition to, and engage in, self-management and adult HIV care and treatment. The specific aims of the study are to:

AIM 1) Assess the impact of a peer mentoring approach to implementing the AIDSTAR-One toolkit on viral suppression and other HIV-related outcomes such as retention in care and adherence to combination antiretroviral therapy (cART), among transitioning youth in different care facility settings (e.g., pediatric hospital, adult hospital, and primary care facilities). Hypothesis: Youth in the intervention arm will experience greater HIV viral suppression at the end of six months of the intervention than youth in the comparison arm.

AIM 1a) Conduct a stratified analysis to examine the impact of a peer mentoring approach separately among: a) the 144 youth participants (15-24) transitioning out of an adolescent clinic into an adult clinic; and b) among 144 youth participants (15-24) who are already attending adult care. This will be a sub-analysis of the larger study to determine the effects of the intervention among these two distinct groups of adolescents and youth.

AIM 2) Examine the experiences of youth and their families, health care providers, peer mentors, and study staff with the peer-mentoring/toolkit program: This objective will be achieved by conducting about 80 qualitative in-depth interviews (IDIs) with the youth participants, as well as about 30 IDIs with their family caregivers. The study team will also interview the health care providers and peer mentors involved in implementing the program, estimated to be around 10 and 12 people respectively. The interviewers will further interview study staff involved in implementing the referral process established for the study (see Section 7.4), estimated to be around 6 people. Out of the 80 youth who will be interviewed, half will be sampled on viral load (VL) test results (e.g. have VL failure at baseline and suppression at midline) and half will be sampled based on VL test results and varying experiences of violence. Interviews with the youth, caregivers, healthcare providers, and peer mentors will provide data on the positive and negative experiences these four groups had with the intervention and the mechanisms believed to support or hinder adolescents' viral suppression. By sampling half of the youth specifically on violence experiences, the study team will also investigate how youth's experiences of violence victimization may relate to their HIV self-management and how the intervention has helped youth deal with these violent experiences, including through the referral procedures established for the study. Interviews with the study staff will offer additional insight into the effectiveness of the referral procedures put in place to support youth with experiences of violence victimization, mental health issues, and other concerns about their wellbeing. These data will contextualize the quantitative data findings and ultimately inform and strengthen the intervention approach.

STUDY DESIGN The study is a randomized controlled trial (RCT) at the individual level. The study team will test a six-month peer-mentoring program among 144 YLHIV in an intervention arm compared to 144 YLHIV in a comparison arm. Participants for the RCT will be consecutively selected from two hospitals -- Arthur Davison Children's Hospital (ADCH) and Ndola Teaching Hospital (NTH) - and two primary care clinics (PCCs) - Twapia Clinic and Lubuto Clinic. The participating facilities were purposively selected because they represent different models of care. ADCH is a hospital for children and serves older youth who should ultimately transition to adult care. In contrast, NTH and the two primary care clinics are essentially adult HIV care settings. While they were not designed to initially serve HIV positive adolescents, they continue to experience a growth in the number of enrolled adolescents. The PCCs were purposively selected based on their high ALHIV patient populations, designated ART center status, and proximity to other study sites.

After the completion of the initial 6-month intervention and the subsequent 6-month follow-up assessment among participants in both arms, the primary intervention group will enter a maintenance phase and the comparison group will receive the intervention for six months. Assessments, including a survey and a blood draw for VL testing, will occur at baseline, at the end of the first six months, and at the end of 12 months. Resistance testing will also be conducted at baseline for those participants who have a VL failure, defined as 1000 copies/ml or higher. Resistance testing is critical for this study as the primary outcome is viral suppression, something that will not occur if a participant has a resistant strain and is not on the correct treatment, no matter how adherent s/he may be. Routine VL results from among ADCH patients reveals that approximately 50% of adolescents have VL failure. Based on that data, it was estimated that 50% of the 288 participants in this research (n=144) will have VL failure and need resistance testing.

At the end of the initial 6-month intervention, study team members will begin conducting qualitative in-depth interviews with participants, their caregivers when possible, and the health care providers, peer mentors, and study staff involved in delivering the program. These data will provide contextual details and experiences to help interpret the study findings and determine what aspects of the intervention were valued.

ELIGIBILITY:
Inclusion Criteria:

* In the age range of 15-24 years
* Aware of her/his HIV status
* On cART for at least six months
* Speaks Bemba or English
* Not planning to move out of the district in the next 18 months
* Planning to be available to attend study activities over the next 18-months, as needed

Exclusion Criteria:

* Being too sick to participate
* Attending boarding school
* Having a sibling already enrolled in the study (one youth per household)
* Having participated in the recent NIH-funded R34 Positive Connections intervention

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 276 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with Viral Suppression (<1000 copies/mL) at Baseline and Midline | ~ 6 months (from baseline to midline)
  <1000 copies/mL

SECONDARY OUTCOMES:
Proportion of Participants with Internalized Stigma (binary, yes to two out of three questions) at baseline and midline. | ~ 6 months (from baseline to midline)
  Internalized stigma was measured at both time points using three agree/disagree questions from the Internalized AIDS Stigma Scale (IA-RSS) (Kalichman et al. AIDSCare 2009). This measure asks participants to either "agree" or "disagree" with each of the following three statements: (1) You feel guilty that you are HIV positive; (2) You are ashamed that you are HIV positive; and (3) You sometimes feel worthless because you are HIV positive to measure self-stigma (also known as internalized stigma). Responses range from 0-3 with 3 indicating higher/worse experiences of internalized stigma. From this data, a binary outcome was generated with "1" indicating that the participant answered "agree" to at least two of the three questions, and "0" otherwise.
Proportion of Participants with Antiretroviral Adherence Treatment Gap at baseline and midline | ~ 6 months (from baseline to midline)
  >= 48 consecutive hours or more of missed ART (self-reported)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Denison, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Arthur Davison Children's Hospital, Ndola, Copperbelt, Zambia

IPD SHARING:
Plan to Share IPD: Yes
The study team plans to share the study data collection tools and de-identified data six months after the study manuscripts are published.
Time Frame: The data will become available six months after the study publications are published.
Access Criteria: Data will be available under Project SOAR's subsection of the Harvard Dataverse repository. Repository link: https://dataverse.harvard.edu/dataverse/projectsoar
URL: https://dataverse.harvard.edu/dataverse/projectsoar

REFERENCES:
- [Background] Amzel A, Toska E, Lovich R, Widyono M, Patel T, Foti C, Dziuban EJ, Phelps BR, Sugandhi N, Mark D, Altschuler J; Child Survival Working Group of the Interagency Task Team on the Prevention and Treatment of HIV-infection in Pregnant Women, Mothers and Children. Promoting a combination approach to paediatric HIV psychosocial support. AIDS. 2013 Nov;27 Suppl 2(0 2):S147-57. doi: 10.1097/QAD.0000000000000098. PMID 24361624
- [Background] Sawyer SM, Drew S, Yeo MS, Britto MT. Adolescents with a chronic condition: challenges living, challenges treating. Lancet. 2007 Apr 28;369(9571):1481-1489. doi: 10.1016/S0140-6736(07)60370-5. PMID 17467519
- [Background] Rosen DS, Blum RW, Britto M, Sawyer SM, Siegel DM; Society for Adolescent Medicine. Transition to adult health care for adolescents and young adults with chronic conditions: position paper of the Society for Adolescent Medicine. J Adolesc Health. 2003 Oct;33(4):309-11. doi: 10.1016/s1054-139x(03)00208-8. No abstract available. PMID 14519573
- [Background] Hussen SA, Chahroudi A, Boylan A, Camacho-Gonzalez AF, Hackett S, Chakraborty R. Transition of youth living with HIV from pediatric to adult-oriented healthcare: a review of the literature. Future Virol. 2015;9(10):921-929. doi: 10.2217/fvl.14.73. PMID 25983853
- [Background] Bal MI, Sattoe JN, Roelofs PD, Bal R, van Staa A, Miedema HS. Exploring effectiveness and effective components of self-management interventions for young people with chronic physical conditions: A systematic review. Patient Educ Couns. 2016 Aug;99(8):1293-309. doi: 10.1016/j.pec.2016.02.012. Epub 2016 Mar 3. PMID 26954345
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Sattoe JN, Bal MI, Roelofs PD, Bal R, Miedema HS, van Staa A. Self-management interventions for young people with chronic conditions: A systematic overview. Patient Educ Couns. 2015 Jun;98(6):704-15. doi: 10.1016/j.pec.2015.03.004. Epub 2015 Mar 17. PMID 25819373
- [Background] Futterman D, Shea J, Besser M, Stafford S, Desmond K, Comulada WS, Greco E. Mamekhaya: a pilot study combining a cognitive-behavioral intervention and mentor mothers with PMTCT services in South Africa. AIDS Care. 2010 Sep;22(9):1093-100. doi: 10.1080/09540121003600352. PMID 20824562
- [Background] Denison JA, Tsui S, Bratt J, Torpey K, Weaver MA, Kabaso M. Do peer educators make a difference? An evaluation of a youth-led HIV prevention model in Zambian Schools. Health Educ Res. 2012 Apr;27(2):237-47. doi: 10.1093/her/cyr093. Epub 2011 Oct 10. PMID 21987477
- [Background] Kim MH, Mazenga AC, Yu X, Ahmed S, Paul ME, Kazembe PN, Abrams EJ. High self-reported non-adherence to antiretroviral therapy amongst adolescents living with HIV in Malawi: barriers and associated factors. J Int AIDS Soc. 2017 Mar 30;20(1):21437. doi: 10.7448/IAS.20.1.21437. PMID 28406275
- [Background] Pantelic M, Boyes M, Cluver L, Meinck F. HIV, violence, blame and shame: pathways of risk to internalized HIV stigma among South African adolescents living with HIV. J Int AIDS Soc. 2017 Aug 21;20(1):21771. doi: 10.7448/IAS.20.1.21771. PMID 28853517
- [Background] Dow DE, Turner EL, Shayo AM, Mmbaga B, Cunningham CK, O'Donnell K. Evaluating mental health difficulties and associated outcomes among HIV-positive adolescents in Tanzania. AIDS Care. 2016 Jul;28(7):825-33. doi: 10.1080/09540121.2016.1139043. Epub 2016 Feb 3. PMID 26837437
- [Background] Woollett N, Cluver L, Bandeira M, Brahmbhatt H. Identifying risks for mental health problems in HIV positive adolescents accessing HIV treatment in Johannesburg. J Child Adolesc Ment Health. 2017 May;29(1):11-26. doi: 10.2989/17280583.2017.1283320. Epub 2017 Mar 13. PMID 28287023
- [Background] Gari T, Habte D, Markos E. HIV positive status disclosure among women attending art clinic at Hawassa University Referral Hospital, South Ethiopia. East Afr J Public Health. 2010 Mar;7(1):87-91. PMID 21413581
- [Background] Maeri I, El Ayadi A, Getahun M, Charlebois E, Akatukwasa C, Tumwebaze D, Itiakorit H, Owino L, Kwarisiima D, Ssemmondo E, Sang N, Kabami J, Clark TD, Petersen M, Cohen CR, Bukusi EA, Kamya M, Havlir D, Camlin CS; SEARCH Collaboration. "How can I tell?" Consequences of HIV status disclosure among couples in eastern African communities in the context of an ongoing HIV "test-and-treat" trial. AIDS Care. 2016;28 Suppl 3(Suppl 3):59-66. doi: 10.1080/09540121.2016.1168917. PMID 27421052
- [Background] Watt MH, Dennis AC, Choi KW, Ciya N, Joska JA, Robertson C, Sikkema KJ. Impact of Sexual Trauma on HIV Care Engagement: Perspectives of Female Patients with Trauma Histories in Cape Town, South Africa. AIDS Behav. 2017 Nov;21(11):3209-3218. doi: 10.1007/s10461-016-1617-1. PMID 27866288
- [Background] Iliyasu Z, Abubakar IS, Babashani M, Galadanci HS. Domestic violence among women living with HIV/AIDS in Kano, Northern Nigeria. Afr J Reprod Health. 2011 Sep;15(3):41-9. PMID 22574491
- [Background] Hatcher AM, Turan JM, Leslie HH, Kanya LW, Kwena Z, Johnson MO, Shade SB, Bukusi EA, Doyen A, Cohen CR. Predictors of linkage to care following community-based HIV counseling and testing in rural Kenya. AIDS Behav. 2012 Jul;16(5):1295-307. doi: 10.1007/s10461-011-0065-1. PMID 22020756
- [Background] Lichtenstein B. Domestic violence in barriers to health care for HIV-positive women. AIDS Patient Care STDS. 2006 Feb;20(2):122-32. doi: 10.1089/apc.2006.20.122. PMID 16475893
- [Background] Hatcher AM, Smout EM, Turan JM, Christofides N, Stockl H. Intimate partner violence and engagement in HIV care and treatment among women: a systematic review and meta-analysis. AIDS. 2015 Oct 23;29(16):2183-94. doi: 10.1097/QAD.0000000000000842. PMID 26353027
- [Derived] Merrill KG, Campbell JC, Kennedy CE, Burke VM, Miti S, Frimpong C, Decker MR, Abrams EA, Mwansa JK, Denison JA. 'So hurt and broken': A qualitative study of experiences of violence and HIV outcomes among Zambian youth living with HIV. Glob Public Health. 2022 Mar;17(3):444-456. doi: 10.1080/17441692.2020.1864749. Epub 2021 Jan 11. PMID 33428559
- [Derived] Denison JA, Burke VM, Miti S, Nonyane BAS, Frimpong C, Merrill KG, Abrams EA, Mwansa JK. Project YES! Youth Engaging for Success: A randomized controlled trial assessing the impact of a clinic-based peer mentoring program on viral suppression, adherence and internalized stigma among HIV-positive youth (15-24 years) in Ndola, Zambia. PLoS One. 2020 Apr 2;15(4):e0230703. doi: 10.1371/journal.pone.0230703. eCollection 2020. PMID 32240186